CLINICAL TRIAL: NCT04242394
Title: If Chronic Gallbladder Diseases Increase the Occurence of Post Endoscopic Retrograde Choledochopancreatography Choledocholithiasis（a Prospective Multi-center Cohort Study)
Brief Title: If Chronic Gallbladder Diseases Increase the Incidence of PEC
Status: Completed | Type: Observational
Sponsor: Hepatopancreatobiliary Surgery Institute of Gansu Province (Other)
Responsible Party: Principal Investigator, Wenbo Meng, M.D., Ph. D, Direct of surgery, Hepatopancreatobiliary Surgery Institute of Gansu Province
Other Study IDs: Chronic gallbladder disease
Record Dates: First submitted 2020-01-22; First posted 2020-01-27 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Cholecystitis
Keywords: ERCP; Acute purulent cholecystitis; Bile duct stone; Post-ERCP-Choledocholithiasis PEC
MeSH Terms: conditions — Cholecystitis; Cholecystolithiasis | interventions — Cholangiopancreatography, Endoscopic Retrograde

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Chronic gallbladder diseases: Routine ERCP participants with chronic gallbladder diseases
  Interventions: Procedure: ERCP
- Without Chronic gallbladder disease: Routine ERCP participants without chronic gallbladder diseases
  Interventions: Procedure: ERCP

INTERVENTIONS:
Procedure: ERCP — Routine ERCP procedures with gallbladder in situ patient

SUMMARY:
This is a prospective, multi-centre trial conducts at 4 ERCP centers in China designed to determine if chronic gallbladder diseases increase the incidence of Post-Endoscopic Retrograde Choledochopancreatography-Choledocholithiasis (PEC)

DETAILED DESCRIPTION:
Endoscopic Retrograde Choledochopancreatography(ERCP) has the advantages of less injury and faster recovery for common bile duct stone patients. However, according to our retrospective study, ERCP will has a mostly 10% possibility to get an acute purulent cholecystitis which often requires emergency intervention, when patients combined with chronic gallbladder diseases, such as chronic cholecystitis, asymptomatic gallstones, and gallbladder wall thickness, the incidence of PEC will increase accordingly. The aim of this study is to observe if chronic gallbladder disease will increase the occurence of PEC and develop a high-risk PEC model.

ELIGIBILITY:
Inclusion Criteria:

* ERCP patients with gallbladder in situ

Exclusion Criteria:

* Acute cholecystitis before surgery
* Gallbladder has been removed
* Gastrointestinal reconstruction
* Unwillingness or inability to consent for the study
* Unstable vital signs Coagulation dysfunction (INR>1.5)
* Low peripheral blood platelet count (<50×10 ^9 / L) or using anti-coagulation drugs
* Preoperative coexistent diseases: acute pancreatitis, GI tract hemorrhage, severe liver disease (such as decompensated liver cirrhosis, liver failure and so on), septic shock Biliary- duodenal fistula confirmed during ERCP
* Pregnant women or breastfeeding

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Common bile duct stone ERCP patients with gallbladder in situ
Sampling Method: Probability Sample
Enrollment: 1019 (Actual)
Dates: Start 2020-02-14 (Actual); Primary Completion 2024-11-16 (Actual); Study Completion 2024-11-16 (Actual)

PRIMARY OUTCOMES:
Number of Acute PEC(post-ERCP-cholecystitis ) | 1month
  When the PEC occurs, with right upper abdominal pain, White Blood Cell increasing, gallbladder wall ≥4mm or crudely, temperature might be more than 38 degree centigrade

SECONDARY OUTCOMES:
Number of Pancreatitis | 1month
  Typical abdominal pain, with the level of serum amylase increasing at least 3 times of the normal range within 24 hours after ERCP.
Number of Cholangitis | 1 month
  Temperature should be more than 38 #, right upper abdominal pain, chills or WBC≥10
Number of Perforation | 1 month
  Typical abdominal pain,abdominal muscle tension, tenderness, evidence of free gas in abdominal cavity

CONTACTS AND LOCATIONS:
Overall Officials: Wenbo Meng, M.D., Ph. D., Principal Investigator — Hepatopancreatobiliary Surgery Institute of Gansu Province
Locations (3):
- China (3):
  - Chinese herb medicine hospital of Longnan City, Longnan, Gansu
  - The first hospital of Tianshui, Tianshui, Gansu
  - Wuwei turmour hospital, Wuwei, Gansu

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cao J, Ding X, Wu H, Shen Y, Zheng R, Peng C, Wang L, Zou X. Classification of the cystic duct patterns and endoscopic transpapillary cannulation of the gallbladder to prevent post-ERCP cholecystitis. BMC Gastroenterol. 2019 Aug 5;19(1):139. doi: 10.1186/s12876-019-1053-6. PMID 31382888
- [Background] Cao J, Peng C, Ding X, Shen Y, Wu H, Zheng R, Wang L, Zou X. Risk factors for post-ERCP cholecystitis: a single-center retrospective study. BMC Gastroenterol. 2018 Aug 22;18(1):128. doi: 10.1186/s12876-018-0854-3. PMID 30134864
- [Derived] Jin B, Wang Y, Zhang X, Zhao J, He W, Jin K, Liu Z, Zhong R, Ma Y, Dong C, Lin Y, Zhu X, Zhu K, Zhang L, Yue P, Li S, Yuan J, Li X, Meng W. Identifying high-risk patients having ERCP as a day surgery with an online prediction platform: Multicohort validation of a machine learning model. Endosc Int Open. 2025 Dec 16;13:a27331387. doi: 10.1055/a-2733-1387. eCollection 2025. PMID 41567602